CLINICAL TRIAL: NCT01248923
Title: A Study of ARRY-520 and Bortezomib Plus Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-520-111
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma, Plasma Cell Leukemia
Keywords: relapsed multiple myeloma; plasma cell dyscrasia; plasmacytoma; kinesin spindle protein; anti-mitotic
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Paraproteinemias; Plasmacytoma | interventions — filanesib; Bortezomib; Proteasome Inhibitors; Injections, Subcutaneous; Dexamethasone; Steroids; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (3):
- ARRY-520 (Schedule 1) + bortezomib + G-CSF (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous; Drug: Bortezomib, proteasome inhibitor; intravenous or subcutaneous; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous
- ARRY-520 (Schedule 1) + bortezomib + dexamethasone + G-CSF (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous; Drug: Bortezomib, proteasome inhibitor; intravenous or subcutaneous; Drug: Dexamethasone, steroid; oral; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous
- ARRY-520 (Schedule 2) + bortezomib + dexamethasone + G-CSF (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous; Drug: Bortezomib, proteasome inhibitor; intravenous or subcutaneous; Drug: Dexamethasone, steroid; oral; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous

INTERVENTIONS:
Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule.
  Arms: ARRY-520 (Schedule 1) + bortezomib + dexamethasone + G-CSF; ARRY-520 (Schedule 2) + bortezomib + dexamethasone + G-CSF
Drug: Bortezomib, proteasome inhibitor; intravenous or subcutaneous — Part 1: standard of care; Part 2: standard of care determined in Part 1.
  Arms: ARRY-520 (Schedule 1) + bortezomib + dexamethasone + G-CSF; ARRY-520 (Schedule 2) + bortezomib + dexamethasone + G-CSF
Drug: Dexamethasone, steroid; oral — Part 1: standard of care; Part 2: standard of care determined in Part 1.
  Arms: ARRY-520 (Schedule 1) + bortezomib + dexamethasone + G-CSF; ARRY-520 (Schedule 2) + bortezomib + dexamethasone + G-CSF
Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous — Part 1: standard of care; Part 2: standard of care.
  Arms: ARRY-520 (Schedule 1) + bortezomib + dexamethasone + G-CSF; ARRY-520 (Schedule 2) + bortezomib + dexamethasone + G-CSF
Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous — Part 1: multiple dose, escalating
  Arms: ARRY-520 (Schedule 1) + bortezomib + G-CSF
Drug: Bortezomib, proteasome inhibitor; intravenous or subcutaneous — Part 1: standard of care
  Arms: ARRY-520 (Schedule 1) + bortezomib + G-CSF
Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous — Part 1: standard of care
  Arms: ARRY-520 (Schedule 1) + bortezomib + G-CSF

SUMMARY:
This is a Phase 1 study during which patients with relapsed or refractory multiple myeloma (MM) or plasma cell leukemia (PCL) will receive investigational study drug ARRY-520 and bortezomib, with or without dexamethasone, with granulocyte-colony stimulating factor (G-CSF) support.

This study has 2 parts. In the first part, patients will receive increasing doses of study drug (2 dosing schedules will be evaluated) in combination with (1) bortezomib with G-CSF support or (2) bortezomib and dexamethasone with G-CSF support, in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Approximately 45 patients from the US will be enrolled in Part 1 (Active, not recruiting).

In the second part of this study, patients will receive the best dose(s) and schedule(s) of study drug, in combination with bortezomib ± dexamethasone + G-CSF, determined from the first part of the study and will be followed to see what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 42 patients from the US will be enrolled in Part 2 (Active, not recruiting).

ELIGIBILITY:
Key Inclusion Criteria (Part 1 and Part 2):

* Confirmed relapsed or refractory MM (measurable disease) or PCL.
* Prior treatment regimens for Part 1: Patients should have received at least 2 prior treatment regimens. Prior treatment must have included at least one full cycle of a proteasome inhibitor (e.g., bortezomib or carfilzomib) and at least one full cycle of an IMiD (e.g., thalidomide, lenalidomide or pomalidomide).
* Prior treatment regimens for Part 2: Patients should have received 1 to 3 prior treatment regimens. Prior treatment could have included bortezomib only if the disease was not refractory to treatment with bortezomib (refractory defined as documented progression on therapy or within 60 days of completing treatment with bortezomib).
* The disease should have progressed per IMWG criteria during or after the last prior treatment regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Adequate hematology laboratory values without transfusion support and without hematological growth factor support within 2 weeks of screening.
* Adequate liver and renal function.
* Additional criteria exist.

Key Exclusion Criteria (Part 1 and Part 2):

* Primary amyloidosis.
* Peripheral neuropathy ≥ Grade 2 or neuropathy with pain, regardless of grade.
* Concomitant malignancies or previous malignancies with less than a 3-year disease free interval at the time of enrollment (patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or Stage A low grade prostate cancer may enroll irrespective of the time of diagnosis).
* Autologous or allogeneic stem cell or bone marrow transplant within 3 months prior to first dose of study drug.
* Treatment with an investigational medicinal product or device within 28 days prior to first dose of study drug.
* Cytotoxic therapy or monoclonal antibodies within 21 days prior to first dose of study drug.
* Radiotherapy within 21 days prior to first dose of study drug (if the radiation portal covered ≤ 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy).
* Major surgery within 14 days and minor surgery within 7 days prior to first dose of study drug.
* Corticosteroid doses > 10 mg/day of prednisone or equivalent within 14 days prior to first dose of study drug.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or active hepatitis C.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-12; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in combination with bortezomib ± dexamethasone + G-CSF in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 1
Establish the maximum tolerated dose (MTD) of the study drug in combination with bortezomib ± dexamethasone + G-CSF. | Part 1
Assess the efficacy of study drug in combination with bortezomib ± dexamethasone + G-CSF in terms of best overall response | Part 2

SECONDARY OUTCOMES:
Assess the efficacy of study drug in combination with bortezomib ± dexamethasone + G-CSF in terms of duration of response, time to progression, treatment-free interval and time to next treatment. | Part 1 and Part 2
Characterize the safety profile of the study drug in combination with bortezomib ± dexamethasone + G-CSF in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 2
Assess the pharmacokinetic (PK) drug interactions between ARRY-520 and bortezomib in terms of plasma concentration-time profiles. | Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - City of Hope, Duarte, California
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Associates in Oncology/Hematology, Rockville, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - NYU Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center at Dallas, Dallas, Texas